CLINICAL TRIAL: NCT06870617
Title: Practical Geriatric Assessment (PGA) Implementation Strategies and Correlative Evaluations for Older Adults With Cancer (PACE-70): A Hybrid Implementation-effectiveness Study
Brief Title: Practical Geriatric Assessment (PGA) Implementation Strategies and Correlative Evaluations (PACE-70)
Acronym: PACE-70
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: UPCC 19924
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: Geriatric Assessment; Advanced Cancer; Toxicity
Keywords: PACE-70; Practical geriatric assessment; body composition in cancer; step count in cancer; Start low go slow
MeSH Terms: interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PGA Implementation Cohort (n=150): All eligible patients will be evaluated on their completion rates of the practical geriatric assessment.
  Interventions: Other: Practical Geriatric Assessment
- Correlative analyses cohort (n=100)
  Interventions: Other: Practical Geriatric Assessment; Other: Correlation of body composition PGA and step count with outcomes

INTERVENTIONS:
Other: Practical Geriatric Assessment — The PGA will be administered via the electronic health record (EHR), available for patients to complete independently prior to an initial medical oncology visit, or during the visit with staff assistance. Results from the PGA will be shared automatically with clinical teams via the EHR, including a Best Practice Alert highlighting any identified geriatric impairment(s) and ASCO's recommendation for PGA-adapted care.
Other: Correlation of body composition PGA and step count with outcomes — Monitoring of step counts (measured via FitBit) and body composition (measured via standard abdominal CT scans)
  Groups: Correlative analyses cohort (n=100)

SUMMARY:
The use of a geriatric assessment to inform oncologic care for older persons with cancer is an evidence-based practice that improves patient-clinician communication, reduces treatment-related toxicity, and is recommended by national guidelines. However, the implementation of a geriatric assessment can be time-consuming and burdensome, leading to suboptimal use in clinical practice. Developed and endorsed by the American Society for Clinical Oncology (ASCO), the Practical Geriatric Assessment (PGA) is designed to improve clinical usability and adoption, but its implementation in real-world settings has not been evaluated. The PACE-70 study aims to evaluate PGA implementation and resultant chemotherapy dose modification among older adults with advanced cancer treated in a community setting. An exploratory aim will evaluate how the PGA, body composition (via abdominal computed tomography scan) and step count monitoring (via FitBit) correlate with chemotherapy toxicity and other clinical outcomes.

DETAILED DESCRIPTION:
Advancing age is the most significant risk factor for cancer. By 2040, it is projected that 60 percent of newly diagnosed cancer cases will occur in individuals aged 70 years or older.5 Managing cancer in older adults requires careful evaluation of treatment risks and benefits, as over 70 percent of older patients experience grade 3+ adverse events, which can impact quality of life and necessitate therapy modifications.6 Moreover, adults over 75 years represent less than 2 percent of participants in phase 3 oncology trials despite constituting 20 percent of incident cancer diagnoses. Consequently, the results of these trials which often lead to drug approvals may not generalize to older adult populations, particularly with respect to drug safety and effectiveness.7,8 There is critical need to generate knowledge regarding best practices for oncologic care tailored to older adult populations.

The use of a geriatric assessment to inform oncologic care for older persons with cancer is an evidence-based practice that improves patient-clinician communication, reduces treatment-related toxicity, and is recommended by national guidelines. The American Society of Clinical Oncology (ASCO) recommends the use of a geriatric assessment (GA) for all adults older than 65 years, and GA-guided management among those with identified impairment. GA-guided management strategies include using GA results to inform cancer treatment decision-making (ie, with respect to treatment selection and/or dose modification) and to address impairments through appropriate interventions, counseling, and referrals.9,10

Despite these recommendations, geriatric assessment is infrequently used in routine practice. Studies have shown that the majority (80 percent) of oncologists do not use a formal geriatric assessment to inform treatment decisions for their older patients. Developed by ASCO, the Practical Geriatric Assessment (PGA) is a novel, validated, pragmatic method of geriatric assessment that relies heavily on patient and caregiver-reported information. It was developed in response to the perception of the comprehensive geriatric assessment as "too cumbersome to incorporate into routine practice" (44%) or "adding no value" (36%). 11 While PGA holds promise for increasing adoption of geriatric assessment in routine oncology care, its feasibility and real-world implementation remain poorly understood, particularly in community oncology settings where most older adults receive care.

The PACE-70 study aims to evaluate novel implementation strategies for the PGA in routine clinical practice for older adults with cancer treated in a community setting. The primary objective is to assess rates of PGA completion. The secondary objective is to evaluate how PGA findings influence dose modification of anti-cancer therapy. Additionally, this trial will explore associations between PGA findings, body composition, and step count monitoring with chemotherapy toxicity and other clinical outcomes. This exploratory aim seeks to determine whether integrating digital technologies with PGA can better predict vulnerability and guide personalized care in older adults with cancer.

The PACE-70 study is a Type III hybrid implementation-effectiveness study enrolling at three community sites within a large academic health system. Eligible participants will be 70 years or older, have a diagnosis of advanced or metastatic solid malignancy, and be starting a new line of palliative-intent systemic therapy, where the expected prevalence of grade 3 toxicity exceeds 50 percent. The PGA will be administered via the electronic health record (EHR), available for patients to complete independently prior to an initial medical oncology visit, or during the visit with staff assistance. Results from the PGA will be shared automatically with clinical teams via the EHR, including a Best Practice Alert highlighting any identified geriatric impairment(s) and ASCO's recommendation for PGA-adapted care. The primary outcome will be the PGA completion rate. The secondary outcome will be the rate of chemotherapy dose modification among those with any identified geriatric impairment. Clinician perspectives on PGA implementation will be assessed via structured interviews among a sub-sample of participating clinicians. In a subsample of patients consenting to additional data collection, exploratory analyses will examine correlations between the PGA, step counts (measured via FitBit) and body composition (measured via standard abdominal CT scans) with clinical outcomes, including toxicity, hospitalization, and death.

ELIGIBILITY:
For PGA Implementation Cohort, patients must meet the following criteria:

1. Age greater than or equal to 70 years.
2. Diagnosis of advanced or metastatic solid malignancy
3. Initiating a new line of palliative-intent systemic therapy with a prevalence of grade 3 toxicity exceeding 50%.

For Correlative Analysis Cohort, patients must additionally meet the following criteria:

1. Must read and speak English and be able to fill out surveys
2. Ability to walk independently or with the use of an assistive device (e.g., walker, cane)
3. Consents to participate in correlative analysis cohort with Fitbit monitoring, body composition analysis, and self-report surveys
4. Have a smartphone able to operate with the Fitbit

For PGA Implementation Cohort, there are no specific exclusion criteria other than not meeting inclusion criteria.

For Correlative Analysis Cohort, patients will be excluded if meeting any of the following criteria:

1. Unable to effectively read and speak English
2. Reliance on a wheelchair, ECOG of 3 or above, clinically bedbound, or unable to walk without assistance every day for the past 7 days (ECOG 3 is confined to bed or chair for more than 50% of waking hours)
3. Concurrent enrollment in a therapeutic clinical trial (as clinical trials often have a substantial symptom-reporting structure). Non-therapeutic clinical trial enrollment is permitted
4. Lack of clinician consent to approach patient

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible participants will be 70 years or older, have a diagnosis of advanced or metastatic solid malignancy, and be starting a new line of palliative-intent systemic therapy, where the expected prevalence of grade 3 toxicity exceeds 50 percent.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Implementation of the PGA | 14 days of initial oncology visit
  The proportion of eligible patients with a completed geriatric assessment within 14 days of initial oncology visit.

SECONDARY OUTCOMES:
Rates of dose modification | Prior to cycle 1 of systemic chemotherapy.
  The proportion of patients with geriatric impairment whose initial cycle of systemic therapy is dose modified.

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Sedhom, M.D., Principal Investigator — Penn Princeton; Samuel Takvorian, M.D., Principal Investigator — Abramson Cancer Center
Locations (3):
- United States (3):
  - Penn Medicine Princeton Medical Center, Princeton, New Jersey
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dale W, Williams GR, R MacKenzie A, Soto-Perez-de-Celis E, Maggiore RJ, Merrill JK, Katta S, Smith KT, Klepin HD. How Is Geriatric Assessment Used in Clinical Practice for Older Adults With Cancer? A Survey of Cancer Providers by the American Society of Clinical Oncology. JCO Oncol Pract. 2021 Jun;17(6):336-344. doi: 10.1200/OP.20.00442. Epub 2020 Oct 15. PMID 33064058
- [Background] Dale W, Klepin HD, Williams GR, Alibhai SMH, Bergerot C, Brintzenhofeszoc K, Hopkins JO, Jhawer MP, Katheria V, Loh KP, Lowenstein LM, McKoy JM, Noronha V, Phillips T, Rosko AE, Ruegg T, Schiaffino MK, Simmons JF Jr, Subbiah I, Tew WP, Webb TL, Whitehead M, Somerfield MR, Mohile SG. Practical Assessment and Management of Vulnerabilities in Older Patients Receiving Systemic Cancer Therapy: ASCO Guideline Update. J Clin Oncol. 2023 Sep 10;41(26):4293-4312. doi: 10.1200/JCO.23.00933. Epub 2023 Jul 17. PMID 37459573
- [Background] Williams GR, Hopkins JO, Klepin HD, Lowenstein LM, Mackenzie A, Mohile SG, Somerfield MR, Dale W. Practical Assessment and Management of Vulnerabilities in Older Patients Receiving Systemic Cancer Therapy: ASCO Guideline Questions and Answers. JCO Oncol Pract. 2023 Sep;19(9):718-723. doi: 10.1200/OP.23.00263. Epub 2023 Jul 17. No abstract available. PMID 37459585
- [Background] Green AK, Tabatabai SM, Aghajanian C, Landgren O, Riely GJ, Sabbatini P, Bach PB, Begg CB, Lipitz-Snyderman A, Mailankody S. Clinical Trial Participation Among Older Adult Medicare Fee-for-Service Beneficiaries With Cancer. JAMA Oncol. 2022 Dec 1;8(12):1786-1792. doi: 10.1001/jamaoncol.2022.5020. PMID 36301585
- [Background] Mohile SG, Mohamed MR, Xu H, Culakova E, Loh KP, Magnuson A, Flannery MA, Obrecht S, Gilmore N, Ramsdale E, Dunne RF, Wildes T, Plumb S, Patil A, Wells M, Lowenstein L, Janelsins M, Mustian K, Hopkins JO, Berenberg J, Anthony N, Dale W. Evaluation of geriatric assessment and management on the toxic effects of cancer treatment (GAP70+): a cluster-randomised study. Lancet. 2021 Nov 20;398(10314):1894-1904. doi: 10.1016/S0140-6736(21)01789-X. Epub 2021 Nov 3. PMID 34741815
- [Background] Versteeg KS, Konings IR, Lagaay AM, van de Loosdrecht AA, Verheul HMW. Prediction of treatment-related toxicity and outcome with geriatric assessment in elderly patients with solid malignancies treated with chemotherapy: a systematic review. Ann Oncol. 2014 Oct;25(10):1914-1918. doi: 10.1093/annonc/mdu052. Epub 2014 Feb 25. PMID 24569912
- [Background] Garner WB, Smith BD, Ludmir EB, Wakefield DV, Shabason J, Williams GR, Martin MY, Wang Y, Ballo MT, VanderWalde NA. Predicting future cancer incidence by age, race, ethnicity, and sex. J Geriatr Oncol. 2023 Jan;14(1):101393. doi: 10.1016/j.jgo.2022.10.008. Epub 2022 Oct 28. PMID 36692964